CLINICAL TRIAL: NCT05003973
Title: The Effectiveness of Anti-resistance Exercise on Lower Limb Lymphoedema Among Gynecological Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Yu-Yun Hsu, Professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-ER-107-433
Record Dates: First submitted 2021-07-26; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Gynecological Cancer; Lower Limb Lymphedema
Keywords: Women's Health; Home-based Anti-Resistance Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- home-based anti-resistance exercise (Experimental)
  Interventions: Behavioral: home-based anti-resistance exercise; Behavioral: usually care
- usually care (Experimental)
  Interventions: Behavioral: usually care

INTERVENTIONS:
Behavioral: home-based anti-resistance exercise — It is a 12-week, middle-level, home-based, anti-resistance exercise. Exercise was recommended 1-2 times per day for 15-20 mins per session.
  Arms: home-based anti-resistance exercise
Behavioral: usually care — The leaflet of the lymphedema self-care, including skin care and manual lymphatic drainage

SUMMARY:
Background:

The incidence of lower limb lymphedema (LLL) after gynecological cancer surgery with lymphadenectomy is about 10-46%. Lower limb lymphedema results in limited physical mobility and reduced patients' quality of life. A hospital -based complete decongestive therapy has been recommended to patients with LLL, including exercise, manual lymphatic drainage, compression therapy, and skin care. However, the inconvenience of the hospital-based rehabilitation program limit the availability for those patients LLL. Home-based exercise program may be feasible instead of the hospital-based program. Few studies have evaluated the effectiveness of the home-based lower extremity exercise on reliving LLL and improving quality of life in patients with LLL.

Research Purposes:

The main purpose of the study is to evaluate the effectiveness of a home-based exercise program for relieving lower extremity lymphedema, including circumference measurement, bioimpedance spectroscopy (BIS), lower limb muscle strength, quality of life related to cancer & LLL, and fatigue.

Methods:

This study is a two- year project with a single-blind randomized clinical trial. The participants are women with gynecological cancer surgery, aged of 20-75 years and currently have lower extremity lymphedema. A sample of 76 participants will be stratified randomly assigned to an experimental group or a control group. The experimental group is to carry out a home-based anti-resistance exercise with elastic band other than a routine care of complex decongestive physiotherapy; while the control group is to carry out a routine care of complex decongestive physiotherapy. The home-based program is a 12-week exercise program. Data collections will be conducted before exercise (Baseline), during exercise (second months), and exercise program after completion. Measures includes (1) Physical examination: limb leg circumference measurement, bioimpedance spectroscopy (BIS), lower limb muscle strength, (2) Questionnaires: Functional status of lymphatic edema of LLL, fatigue, and EORTC-QLQ-C30.

Anticipated Outcomes:

Findings from this study could provide a reference of home-based exercise guideline and be integrated into the care of activities for women following gynecological surgery with LLL.

ELIGIBILITY:
Inclusion Criteria:

* women with gynecological cancer surgery
* aged of 20-75 years
* currently have lower extremity lymphedema.

Exclusion Criteria:

* heart failure
* kidney failure
* DVT
* limb surgery

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-20 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Limb circumference change from baseline to 3 months | from baseline to 3 months
  Measuring by measuring tape
Edema change from baseline to 3 months | from baseline to 3 months
  Measuring by Bioelectrical Impedance Spectroscopy (BIS)- InBody S10
Lower limb muscle strength change from baseline to 3 months | from baseline to 3 months
  Measuring by microFET 2
Functional status of lymphatic edema of LLL change from baseline to 3 months | from baseline to 3 months
  Measuring by Lymphoedema Functioning, Disability and Health Questionnaire for Lower Limb Lymphoedema (Lymph-ICF-LL). It is a 28-item, 0(no problem) to 10(very severe) questionnaire.
Fatigue change from baseline to 3 months | from baseline to 3 months
  Measuring by Chinese Lee Fatigue Scale Short Form (C-LESSF). It is a 7-item, from 0(no fatigue) to 10(very fatigue) questionnaire.
EORTC-QLQ-C30 | from baseline to 3 months
  Measuring by EORTC QLQ C30. It is a 30-item, from 0(no problem) to 10(very severe) questionnaire.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939